CLINICAL TRIAL: NCT00617916
Title: Hyperspectral Imaging to Assess and Predict Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: HyperMed (Industry)
Collaborators: The Cleveland Clinic (Other); Olive View-UCLA Education & Research Institute (Other); University of Pennsylvania (Other)
Responsible Party: Kevin Schomacker, PhD, HyperMed, Inc.
Other Study IDs: 2005-001; R42DK069871 (NIH)
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Diabetic Foot Ulcers
Keywords: hyperspectral imaging; tissue oxygenation; diabetic foot ulcers; wound healing; prevention
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to test a prototype imaging instrument that relies on Medical HyperSpectral Imaging (MHSI) technology for the assessment and prediction of diabetic foot ulceration and wound healing. The imaging system utilizes the biomarkers of oxyhemoglobin (oxyHb) and deoxyhemoglobin (deoxyHb), in the upper layers of skin on the foot as: a metric for assessing wound healing, a reflection of microvascular disease, and determining tissue at risk for forming new ulcers. MHSI results will also be compare with ABI and TcPO2 measurements.

DETAILED DESCRIPTION:
ULCER HEALING STUDY: This is a study comparing measurements from a cohort of 66 diabetic subjects (30 Type 1 and 36 Type 2) with at least one foot ulcer. The study will take place at three medical centers. Each center will enroll 22 subjects (10 Type 1 and 12 Type 2). Subjects will be required to participate in eleven (11) clinic visits over a 6 month period. The first visit will last approximately three hours and each of the other visits will last about two hours. The eleven visits will be scheduled as follows in the Table to the right.

At the initial visit the subject will give informed consent and a full medical history, and will schedule the dates of the remaining visits for the study. The subject recruiter will contact each subject one week prior to each subsequent visit to either confirm the subject's attendance or to re-schedule the visit.

NEW ULCER PREDICTION STUDY: This is a study comparing measurements of 210 "high risk" diabetic subjects (90 Type 1 and 120 Type 2) over an 18-24 month period. The study will take place at three medical centers. Each center will enroll 70 subjects (30 Type 1 and 40 Type 2). Subjects will all be required to participate in nine (9) clinic visits. The nine visits will be scheduled as follows in the Table to the right.

The first visit will last approximately three hours and each of the other visits will last about 2 hours. At the initial visit the subject will give informed consent and a full medical history, and will schedule the dates of the visits for the rest of the study. The subject recruiter will contact each subject one week prior to each subsequent visit to either confirm the subject's attendance or to re-schedule the visit.

ELIGIBILITY:
Ulcer Healing Study

Inclusion Criteria:

* Subjects with Type 1 diabetes (defined as diabetes beginning before age 35, requiring insulin, and diagnosed with diabetes for more than six months) or Type 2 diabetes.
* Presence of at least one foot ulcer

Exclusion criteria:

* Peripheral arterial occlusive disease (PAD) that is severe enough to require surgical bypass operation.
* Cardiovascular disease as demonstrated in only these instances: congestive heart failure that leads to severe edema at the lower extremity, stroke or transient ischemic attack with residual nerve dysfunction.
* Uncontrolled hypertension: SBP>190 mmHg or DBP > 110 mmHg
* End stage renal disease (subjects on renal dialysis or kidney transplantation)
* Any other serious chronic disease that can affect wound healing
* Subjects currently on any of the following medications: Glucocorticoids, Antineoplastics
* Females if lactating or pregnant or, if of childbearing potential, unwilling to use standard birth control. All females of childbearing potential will undergo a pregnancy test during each visit.

NEW ULCER PREDICTION STUDY:

Inclusion criteria:

* Subjects with Type 1 diabetes (defined as diabetes beginning before age 35, requiring insulin, and diagnosed with diabetes for more than six months) or Type 2 diabetes.
* Subject without foot ulcers but at "high risk" for foot ulceration. In order to define "high risk" for this study, we are using the International Working Group standards:

  1. Advanced neuropathy, defined by loss of protective sensation in the foot with a vibrational perception threshold (VPT) over 25mHz or inability to detect Semmes Weinstein 5.07 (10g) monofilament
  2. Presence of significant deformity
  3. Peripheral vascular disease with ankle brachial index < 0.7
  4. History of previous ulceration or presence of a foot ulcer
  5. At least one foot that is ulcer free at the time of enrollment

Exclusion criteria:

* Peripheral arterial occlusive disease (PAD) that is severe enough to require surgical bypass operation.
* Cardiovascular disease as demonstrated in only these instances: congestive heart failure that leads to severe edema at the lower extremity, stroke or transient ischemic attack with residual nerve dysfunction.
* Uncontrolled hypertension: SBP > 190 mmHg or DBP > 110 mmHg
* End stage renal disease (subjects on renal dialysis or kidney transplantation)
* Any other serious chronic disease that can affect wound healing
* Subjects on any of the following medications: Glucocorticoids and Antineoplastic agents
* Females if lactating or pregnant or, if of childbearing potential, unwilling to use standard birth control. All females of childbearing potential will undergo a pregnancy test during each visit.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic population - diabetic patients at high risk for ulceration
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Davis, PhD, Principal Investigator — The Cleveland Clinic; Aksone Nouvong, DPM, Principal Investigator — Olive View-UCLA Education & Research Institute; Emile Mohler, MD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Olive View UCLA Medical Center, Sylmar, California
  - Lerner Research Institute, The Cleveland Clinic, Cleveland, Ohio
  - University of Pennslyvania Healthcare System, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Greenman RL, Panasyuk S, Wang X, Lyons TE, Dinh T, Longoria L, Giurini JM, Freeman J, Khaodhiar L, Veves A. Early changes in the skin microcirculation and muscle metabolism of the diabetic foot. Lancet. 2005 Nov 12;366(9498):1711-7. doi: 10.1016/S0140-6736(05)67696-9. PMID 16291064
- [Background] Cancio LC, Batchinsky AI, Mansfield JR, Panasyuk S, Hetz K, Martini D, Jordan BS, Tracey B, Freeman JE. Hyperspectral imaging: a new approach to the diagnosis of hemorrhagic shock. J Trauma. 2006 May;60(5):1087-95. doi: 10.1097/01.ta.0000217357.10617.3d. PMID 16688075
- [Background] Khaodhiar L, Dinh T, Schomacker KT, Panasyuk SV, Freeman JE, Lew R, Vo T, Panasyuk AA, Lima C, Giurini JM, Lyons TE, Veves A. The use of medical hyperspectral technology to evaluate microcirculatory changes in diabetic foot ulcers and to predict clinical outcomes. Diabetes Care. 2007 Apr;30(4):903-10. doi: 10.2337/dc06-2209. Epub 2007 Feb 15. PMID 17303790
- [Background] Panasyuk SV, Yang S, Faller DV, Ngo D, Lew RA, Freeman JE, Rogers AE. Medical hyperspectral imaging to facilitate residual tumor identification during surgery. Cancer Biol Ther. 2007 Mar;6(3):439-46. doi: 10.4161/cbt.6.3.4018. Epub 2007 Mar 16. PMID 17374984
- [Derived] Nouvong A, Hoogwerf B, Mohler E, Davis B, Tajaddini A, Medenilla E. Evaluation of diabetic foot ulcer healing with hyperspectral imaging of oxyhemoglobin and deoxyhemoglobin. Diabetes Care. 2009 Nov;32(11):2056-61. doi: 10.2337/dc08-2246. Epub 2009 Jul 29. PMID 19641161